CLINICAL TRIAL: NCT00823095
Title: The Observational Effects of the Topical Application of ViaNOx-H (Gaseous Nitric Oxide) on the Bio-Burden in Chronic Non-Healing Colonized Ulcers of the Lower Extremities
Brief Title: Topical Nitric Oxide Trial in Chronic Non-Healing Wounds
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Subject recuitment halted and won't resume; subjects are no longer being treated.
Sponsor: Loma Linda University (Other)
Collaborators: Nitric BioTherapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNO-1B; DMF 15551; IND 68617
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Ulcer of Lower Extremity
Keywords: chronic cutaneous ulcers; Nitric Oxide; topically applied; Biofilm; Colonized chronic non-healing ulcers
MeSH Terms: interventions — Nitric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Topically applied Nitric Oxide (Experimental): Topically applied Nitric Oxide for 8 hours daily for 2 weeks.
  Interventions: Drug: Nitric Oxide

INTERVENTIONS:
Drug: Nitric Oxide — Topically applied gaseous nitric oxide at 8 to 10 parts per million, for 8 hours each night for 14 nights.
  Other Names: ViaNOx-H; gaseous nitric oxide; gNO

SUMMARY:
To determine the effects of topically applied ViaNOx-H for 8 hours daily for 2 weeks on the reduction of the bio-burden in biofilms on chronic non-healing wounds as recorded by measurements of wound size and wound culture.

DETAILED DESCRIPTION:
The primary goal of this study is to determine the effects of topically applied gaseous nitric oxide on the bio-burden of chronic non-healing wounds of the lower extremities. Reports will include:

* Comparisons of the demographics and diagnoses of those patients treated with ViaNOx-H.
* Tabulation as to the organisms found and the bio-burden as measured by counts (0 to +4).
* Tabulation of the number and types of adverse events during ViaNOx-H treatment.
* Comparisons of the response of different organisms to ViaNOx-H treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have a chronic (> 8 weeks duration) colonized cutaneous ulcer (defined as a wound containing a local margin of erythema, edema or tenderness; presence of exudates; and/or presence of a malodorous smell)in their lower extremity (below the knee) resulting from either diabetes or venous stasis disease.
* Are 18 years of age or older.

Exclusion Criteria:

* Have had a change in their topical treatment during the last 4 weeks
* Have evidence of Clinical Infection
* Have a transcutaneous oxygen tension <30mmHg
* Have evidence of the ulcer or infection extending to the underlying muscle or bone.
* Are pregnant.
* Are less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takkin Lo, MD, MPH, Principal Investigator — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Topically Applied Nitric Oxide: Topically applied gaseous nitric oxide at 8 to 10 parts per million, for 8 hours each night for 14 nights.
Period: Overall Study
Arm/Group | Topically Applied Nitric Oxide
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Treatment
Arm/Group | Group 1
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 7
Evidence of a colonized wound on the lower extremity. [Number; unit: participants]
  >=65 years | 4
  18 to 65 years | 3

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is the Eradication of the Bio-burden as Measured by a Reduction in Culture Growth to ≤ +2.
Time Frame: at 28 days post enrollment
Population: Data not available for this study due to dissolution of company contracted to perform study analysis
Arm/Group | Group 1
Number analyzed (Participants) | 0

2. Secondary Outcome: The Secondary Endpoint Measure is a Reduction on Wound Size.
Description: reduction in bioburden as assessed by number of cfu's per cm2 on culture
Time Frame: 28 days post enrollment
Population: Data not available for this study due to dissolution of company contracted to perform analysis.
Groups:
- Treatment: reduction in bioburden as assessed by number of cfu's per cm2 on culture
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
No data available for this study due to dissolution of company contracted to perform study analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No